CLINICAL TRIAL: NCT05957588
Title: Non-ventilated Prone Positioning in the COVID-19 Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor St. Luke's Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BaylorSt.Lukes
Record Dates: First submitted 2023-07-07; First posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: COVID-19; Proning; Oxygenation; Length of Stay
Keywords: acute care; self-proning
MeSH Terms: conditions — COVID-19 | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: This study was a prospective randomized cohort study in which data was collected for over 14 days or until discharged to a lower level of care from the telemetry-monitored, acute care unit. Data collected on study participants included the need for escalating respiratory care as well as length of stay in the acute care unit. Comparative analysis was conducted with data collected from hospitalized patients (the control group) with a diagnosis of COVID-19 on a non-ICU acute care, telemetry-monitored unit that met the hypoxemia criteria, but that did not receive the proning intervention. The data from the control group was collected by a retrospective chart analysis after 14 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proning group (Experimental): COVID-19 hypoxemic patients that receive standard of care AND participate in self-proning following the research protocol.
  Interventions: Other: Proning group
- Control group (Other): COVID-19 hypoxemic patients that receive standard of care.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Proning group — Patients were educated about self-proning, and instructed to self-prone every 2 hours. The patient documented their position on the checklists every 2 hours.
  Upon initiation of the initial proning, the patient was monitored by the research team RN for adverse effects for 15 minutes (such as inability to tolerate position or signs of respiratory distress).
  If the patient tolerated the proning well, the RN entered the patient's oxygen saturation into the EMR, and documented the initial position (prone or supine) on the checklist. O2 saturation was documented at least every 4 hours per unit protocol.
  The checklists were placed in a binder at the nurses' station at the end of each shift and collected daily by a member of the research team.
  This intervention for each proned patient continued until either of the following occurred: ei the patient was discharged to a lower level of care or 14 days had passed.
  Arms: Proning group
Other: Control group — A retrospective chart review was completed by the research team to ascertain length of stay, oxygenation, and pressure injuries for the control group on the acute care, telemetry monitored unit.
  Arms: Control group

SUMMARY:
In the COVID-19 healthcare crisis, one possible treatment therapy that has generated the most discussion is that of proning, or the position in which the patient lays face down as opposed to face up for a period of time. As the pandemic continues, this method has been more widely adopted to increase oxygen saturation in patients in respiratory distress. While proning research is both ongoing and extensive in the ICU population of COVID-19 patients, minimal research has been conducted with acute care patients. The researchers aim to address this gap with this study. The researchers used a systematic approach to educate patients and staff about patient self-proning, implementing self-proning every 2 hours, and monitoring escalation of oxygen levels, as well as length of stay in the acute care unit. The researchers hypothesized an improvement in oxygen saturation levels as evidenced by no escalation of respiratory care (i.e. higher levels of oxygen needed, transfer to higher level of care), resulting in shorter lengths of stay for the intervention population.

DETAILED DESCRIPTION:
Background: In the COVID-19 healthcare crisis, one possible treatment therapy that has generated the most discussion is that of proning, or the position in which the patient lays face down as opposed to face up for a period of time. As the pandemic continues, this method has been more widely adopted to aid in increasing oxygen saturation levels in patients in respiratory distress. While proning research is both ongoing and extensive in the ICU population of COVID-19 patients, minimal research has been conducted using acute care patients. The researchers aim to address this gap with this treatment method.

Methods: This study was a randomized controlled trial with a sample size of 216 patients, with 36 self-proners, 104 standard of care patients, and 69 patients refused to participate in the intervention. The researchers also studied rates of attrition for self-proning. Patients were randomized using a randomization table per hospital admission. The researchers consented patients who were oriented, and able to self-prone safely without assistance on an acute care telemetry monitored unit. Patients were self-documenting their position per hour, and the researchers were using the electronic health record to collect vital signs and presence of pressure injuries. All data was entered in the secure REDCap database.

ELIGIBILITY:
Inclusion Criteria:

* patients that were confirmed COVID-19 positive on an acute-care, telemetry-monitored, non-ICU unit and were considered hypoxemic
* conscious, oriented and independently mobile patients
* subjects were patients 18 years and older

Exclusion Criteria:

* negative for COVID 19
* patients in ICU settings
* patients in acute respiratory distress
* patients in hemodynamic instability (systolic blood pressure below 90) or arrhythmia
* patients with altered mental status
* patients with unstable spine/thoracic injury
* patients with recent abdominal surgery
* patients with significant pressure ulcers (above stage 1)
* pregnant patients past the 2nd trimester
* patients that have concerning neurological issues (such as seizures)
* Patients that are unable to change positions independently

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Length of stay | 7 months
  amount of time patient was admitted to acute care unit

SECONDARY OUTCOMES:
Oxygenation | 7 months
  Saturation of partial pressure of oxygen (in Litres)
Pressure injuries | 7 months
  presence skin breakdown using clinically accepted wound staging tool

OTHER OUTCOMES:
demographics | 7 months
  race, ethnicity, height, weight, age, gender

CONTACTS AND LOCATIONS:
Overall Officials: Marie Hodges, BSN, RN, Principal Investigator — Baylor St. Luke's Medical Center
Locations (1):
- Baylor St. Luke's Medical Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Access to trial information can be requested by qualified researchers engaging in independent scientific research and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact geraldine.jones@commonspirit.org; marie.hodges@commonspirit.org; and nishant.varghese@commonspirit.org.
Supporting Information: Study Protocol, ICF
Time Frame: June 2022 - June 2027

REFERENCES:
- [Background] Alser O, Mokhtari A, Naar L, Langeveld K, Breen KA, El Moheb M, Kapoen C, Gaitanidis A, Christensen MA, Maurer LR, Mashbari H, Bankhead-Kendall B, Parks J, Fawley J, Saillant N, Mendoza A, Paranjape C, Fagenholz P, King D, Lee J, Farhat MR, Velmahos GC, Kaafarani HMA. Multisystem outcomes and predictors of mortality in critically ill patients with COVID-19: Demographics and disease acuity matter more than comorbidities or treatment modalities. J Trauma Acute Care Surg. 2021 May 1;90(5):880-890. doi: 10.1097/TA.0000000000003085. PMID 33891572
- [Background] Caputo ND, Strayer RJ, Levitan R. Early Self-Proning in Awake, Non-intubated Patients in the Emergency Department: A Single ED's Experience During the COVID-19 Pandemic. Acad Emerg Med. 2020 May;27(5):375-378. doi: 10.1111/acem.13994. PMID 32320506
- [Background] Cardona S, Downing J, Alfalasi R, Bzhilyanskaya V, Milzman D, Rehan M, Schwartz B, Yardi I, Yazdanpanah F, Tran QK. Intubation rate of patients with hypoxia due to COVID-19 treated with awake proning: A meta-analysis. Am J Emerg Med. 2021 May;43:88-96. doi: 10.1016/j.ajem.2021.01.058. Epub 2021 Jan 27. PMID 33550104
- [Background] Ding L, Wang L, Ma W, He H. Efficacy and safety of early prone positioning combined with HFNC or NIV in moderate to severe ARDS: a multi-center prospective cohort study. Crit Care. 2020 Jan 30;24(1):28. doi: 10.1186/s13054-020-2738-5. PMID 32000806
- [Background] Dubosh NM, Wong ML, Grossestreuer AV, Loo YK, Sanchez LD, Chiu D, Leventhal EL, Ilg A, Donnino MW. Early, awake proning in emergency department patients with COVID-19. Am J Emerg Med. 2021 Aug;46:640-645. doi: 10.1016/j.ajem.2020.11.074. Epub 2020 Dec 3. PMID 33309507
- [Background] Ehrmann S, Li J, Ibarra-Estrada M, Perez Y, Pavlov I, McNicholas B, Roca O, Mirza S, Vines D, Garcia-Salcido R, Aguirre-Avalos G, Trump MW, Nay MA, Dellamonica J, Nseir S, Mogri I, Cosgrave D, Jayaraman D, Masclans JR, Laffey JG, Tavernier E; Awake Prone Positioning Meta-Trial Group. Awake prone positioning for COVID-19 acute hypoxaemic respiratory failure: a randomised, controlled, multinational, open-label meta-trial. Lancet Respir Med. 2021 Dec;9(12):1387-1395. doi: 10.1016/S2213-2600(21)00356-8. Epub 2021 Aug 20. PMID 34425070
- [Background] Garg S, Patel K, Pham H, Whitaker M, O'Halloran A, Milucky J, Anglin O, Kirley PD, Reingold A, Kawasaki B, Herlihy R, Yousey-Hindes K, Maslar A, Anderson EJ, Openo KP, Weigel A, Teno K, Ryan PA, Monroe ML, Reeg L, Kim S, Como-Sabetti K, Bye E, Shrum Davis S, Eisenberg N, Muse A, Barney G, Bennett NM, Felsen CB, Billing L, Shiltz J, Sutton M, Abdullah N, Talbot HK, Schaffner W, Hill M, Chatelain R, Wortham J, Taylor C, Hall A, Fry AM, Kim L, Havers FP. Clinical Trends Among U.S. Adults Hospitalized With COVID-19, March to December 2020 : A Cross-Sectional Study. Ann Intern Med. 2021 Oct;174(10):1409-1419. doi: 10.7326/M21-1991. Epub 2021 Aug 10. PMID 34370517
- [Background] Kallet RH. A Comprehensive Review of Prone Position in ARDS. Respir Care. 2015 Nov;60(11):1660-87. doi: 10.4187/respcare.04271. PMID 26493592
- [Background] McNicholas B, Cosgrave D, Giacomini C, Brennan A, Laffey JG. Prone positioning in COVID-19 acute respiratory failure: just do it? Br J Anaesth. 2020 Oct;125(4):440-443. doi: 10.1016/j.bja.2020.06.003. Epub 2020 Jun 9. No abstract available. PMID 32571573
- [Background] Munshi L, Del Sorbo L, Adhikari NKJ, Hodgson CL, Wunsch H, Meade MO, Uleryk E, Mancebo J, Pesenti A, Ranieri VM, Fan E. Prone Position for Acute Respiratory Distress Syndrome. A Systematic Review and Meta-Analysis. Ann Am Thorac Soc. 2017 Oct;14(Supplement_4):S280-S288. doi: 10.1513/AnnalsATS.201704-343OT. PMID 29068269
- [Background] Qian ET, Gatto CL, Amusina O, Dear ML, Hiser W, Buie R, Kripalani S, Harrell FE Jr, Freundlich RE, Gao Y, Gong W, Hennessy C, Grooms J, Mattingly M, Bellam SK, Burke J, Zakaria A, Vasilevskis EE, Billings FT 4th, Pulley JM, Bernard GR, Lindsell CJ, Rice TW; Vanderbilt Learning Healthcare System Platform Investigators. Assessment of Awake Prone Positioning in Hospitalized Adults With COVID-19: A Nonrandomized Controlled Trial. JAMA Intern Med. 2022 Jun 1;182(6):612-621. doi: 10.1001/jamainternmed.2022.1070. PMID 35435937
- [Background] Rees EM, Nightingale ES, Jafari Y, Waterlow NR, Clifford S, B Pearson CA, Group CW, Jombart T, Procter SR, Knight GM. COVID-19 length of hospital stay: a systematic review and data synthesis. BMC Med. 2020 Sep 3;18(1):270. doi: 10.1186/s12916-020-01726-3. PMID 32878619
- [Background] Taylor SP, Bundy H, Smith WM, Skavroneck S, Taylor B, Kowalkowski MA. Awake Prone Positioning Strategy for Nonintubated Hypoxic Patients with COVID-19: A Pilot Trial with Embedded Implementation Evaluation. Ann Am Thorac Soc. 2021 Aug;18(8):1360-1368. doi: 10.1513/AnnalsATS.202009-1164OC. PMID 33356977
- [Background] Shearer SC, Parsa KM, Newark A, Peesay T, Walsh AR, Fernandez S, Gao WZ, Pierce ML. Facial Pressure Injuries from Prone Positioning in the COVID-19 Era. Laryngoscope. 2021 Jul;131(7):E2139-E2142. doi: 10.1002/lary.29374. Epub 2021 Jan 5. PMID 33389768
- [Background] World Health Organization (WHO). (2020). Clinical management of severe acute respiratory infection when novel coronavirus (nCoV) infection is suspected: Interim guidance. World Health Organization, 1-10. https://www.who.int/publications/i/item/10665-332299
- See also: Enterprise login to find out more about research and innovation — http://commonspirit.org
- Available data/document: Informed Consent Form: Documents — https://irbnet.org/release/study/designer.do?ctx_id=9&spk_id=1793612 — This URL and identifier are used internally by Common Spirit Health IRB. The link is IRBNET.org and registration thru CSH is required. The link provides access to a digital document repository including the consent form.
- Available data/document: Study Protocol: Protocol — https://irbnet.org/release/study/designer.do?ctx_id=9&spk_id=1793612 — This URL and identifier are used internally by Common Spirit Health IRB. The link is IRBNET.org and registration thru CSH is required. The link provides access to a digital document repository including the protocol document.

DOCUMENTS (2):
  • Study Protocol (2023-06-07): https://cdn.clinicaltrials.gov/large-docs/88/NCT05957588/Prot_000.pdf
  • Informed Consent Form (2023-06-07): https://cdn.clinicaltrials.gov/large-docs/88/NCT05957588/ICF_001.pdf